CLINICAL TRIAL: NCT02838355
Title: Employing End Tidal Capnography in Continuous Flow Ventricular Assist Device Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding not received
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Carolyn Miller Reilly, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00082202
Record Dates: First submitted 2016-05-17; First posted 2016-07-20 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Cardiomyopathy; Cardiovascular Disease; Heart Disease
MeSH Terms: conditions — Cardiomyopathies; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Respiration Monitoring (Active Comparator): Participants scheduled for mechanical circulatory support device (MCSD) implant or who have been readmitted to an intensive care unit (ICU) with a continuous flow left ventricular assist device (CF-LVAD) will receive standard respiratory monitoring throughout their stay in the ICU.
  Interventions: Other: Standard Non-invasive Respiratory Depression Monitoring
- Standard Respiration Monitoring + Continuous ETCO2-NC (Experimental): Participants scheduled for mechanical circulatory support device (MCSD) implant or who have been readmitted to an intensive care unit (ICU) with a continuous flow left ventricular assist device (CF-LVAD) will receive standard respiratory monitoring and continuous end-tidal capnography monitoring via nasal cannula (ETCO2-NC) throughout their stay in the ICU.
  Interventions: Device: Respiratory Depression Monitoring with End Tidal Carbon Dioxide Nasal Cannula (ETCO2- NC); Other: Standard Non-invasive Respiratory Depression Monitoring

INTERVENTIONS:
Device: Respiratory Depression Monitoring with End Tidal Carbon Dioxide Nasal Cannula (ETCO2- NC) — The ETCO2-NC is a non-invasive device that monitors the amount of carbon dioxide that is exhaled with every breath.
  Other Names: ETCO2- NC
  Arms: Standard Respiration Monitoring + Continuous ETCO2-NC
Other: Standard Non-invasive Respiratory Depression Monitoring — Standard non-invasive respiration monitoring includes telemetry of heart rate and rhythm, respiratory rate, blood pressure, CF-LVAD flow, and oxygen saturation (SpO2) via pulse oximetry.

SUMMARY:
The purpose of this study is to explore how the End Tidal Carbon Dioxide monitoring via nasal cannula (ETCO2-NC) device may allow for earlier detection of respiratory complications. This device will detect the amount of carbon dioxide exhaled with each breath and may better predict high levels of this than traditional monitoring. This may reduce the number and severity of respiratory issues. A convenience sample of 60 participants either scheduled for continuous flow left ventricular assist device (CF-LVAD) implant or who have been readmitted to an ICU with a CF-LVAD will be recruited and randomized to usual care or usual care plus ETCO2-NC throughout their stay in the ICU.

DETAILED DESCRIPTION:
The purpose of this proposal is to explore the relationships between End Tidal Carbon Dioxide (ETCO2) via nasal cannula (ETCO2-NC) and routinely measured physiologic and participant reported parameters in extubated participants who have received a continuous flow left ventricular assist device (CF-LVAD), and to determine if the addition of ETCO2-NC monitoring to usual care is associated with decreased incidence and severity of respiratory issues.

A convenience sample of 60 participants either scheduled for mechanical circulatory support device (MCSD) implant or who have been readmitted to an intensive care unit (ICU) with a CF-LVAD will be recruited and randomized to usual care or usual care plus ETCO2-NC throughout their stay in the ICU.

Investigators seek to examine the relationship between ETCO2-NC with traditional physiologic measures, clinical assessments, and participant reported symptoms in persons with a CF-LVAD. Additionally, this study intends to compare the respiratory outcomes of extubated persons with a CF-LVAD randomized to usual care to those receiving usual care plus ETCO2- NC.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for mechanical circulatory support device (MCSD) implant or have been readmitted to an intensive care unit (ICU) with a continuous flow left ventricular assist device (CF-LVAD)
* New York Heart Association (NYHA) functional class III to IV
* Ability to read, write, and speak English

Exclusion Criteria:

* Requiring mechanical ventilation during the active phase of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Respiratory Distressed assessed by Respiratory Distress Observation Scale (RDOS) | Up to 2 Weeks
  The RDOS is an ordinal level scale with eight observer-rated parameters: heart rate, respiratory rate, accessory muscle use, paradoxical breathing pattern, restlessness, grunting at end-expiration, nasal flaring, and a fearful facial display. Each parameter is scored from 0 to 2 points and the points are summed. Scale scores range from 0 signifying no distress to 16 signifying the most severe distress.
Dyspnea Rate assessed by the Dyspnea Visual Analogue Scale (DVAS) | Up to 2 Weeks
  The DVAS is a self-reported scale that asks participants to indicate how much shortness of breath they are experiencing by marking on a line 100 mm in length between "no shortness of breath" and "shortness of breath as bad as can be".
Incidence of Respiratory Depression | Up to 2 Weeks
  This is physiologic data abstracted from the medical record: respiration that has a rate below 12 breaths per minute or that fails to provide full ventilation and perfusion of the lungs.
Severity of Respiratory Depression | Up to 2 Weeks
  Physiologic data abstracted from the medical record: Severity of respiration depression will be collected via standard hospital code met and code blue forms. Respiratory compromise will be defined as respiratory rate increase or decrease by 20% or greater, an ETCO2 value greater than 20% above baseline values, or a SpO2 less than 90% for greater than 10 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Reilly, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States